CLINICAL TRIAL: NCT00774540
Title: Acute Pain and Role of Ketolorac in Inflammatory Mediators After Knee Arthroscopy Evaluated by Microdialysis
Brief Title: Acute Pain and Inflammation After Surgery
Acronym: Knemikro01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Leiv Arne Rosseland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Knemikro01; S-04342
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Knee Injuries
Keywords: Acute pain; Inflammatory pain; Inflammatory mediators; Pain relief; Microdialysis
MeSH Terms: conditions — Knee Injuries; Acute Pain | interventions — Ketorolac; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ketorolac
  Interventions: Drug: 1 Ketorolac intraarticular
- 2 (Placebo Comparator): saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1 Ketorolac intraarticular — Ketorolac intraarticular 5 mg
  Other Names: Ketorolac; Saline
  Arms: 1
Drug: Placebo — Saline
  Arms: 2

SUMMARY:
The purpose of this study is

1. to observe acute pain after surgery and measure the natural course of inflammatory mediators
2. study pain relieving effects and local anti-inflammatory effects of systemically administered ketorolac

DETAILED DESCRIPTION:
Randomizized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Day case surgical patients above 18 years old
* Non pregnant

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain relief local anti-flammatory effects | 2 h

SECONDARY OUTCOMES:
Rescue analgesic consumption | 2 h

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Arne Rosseland, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Division of Emergencies and Critical Care, Oslo, Norway